CLINICAL TRIAL: NCT05631392
Title: A Prospective, Non-randomised, Multi-centre, Post-market Clinical Follow-up Observational Study to Evaluate the Clinical and Radiographic Outcomes of the BEE® HA Cage for Anterior Cervical Discectomy and Fusion.
Brief Title: Study to Evaluate the Clinical and Radiographic Outcomes of the BEE® HA Cage for Anterior Cervical Discectomy and Fusion
Status: Recruiting | Type: Observational
Sponsor: Invibio Ltd (Industry)
Collaborators: NGMedical GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: NGM01
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Cervical Disc Degeneration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational data collection of information after undergoing standard Cervical spine fusion surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 years of age or older (≥ 18 years) and are skeletally mature.
2. Subjects with discopathy, disc hernia with radiculopathy and/or myelopathy, or stenosis of the foramen and spinal canal with or without cervical radiculopathy/myelopathy, at one or two contiguous levels from C3 to C7, and confirmed by imaging studies (CT and/or MRI will be taken according to standard local procedures and confirmed by the Investigator that imaging represents the indication for surgery).
3. Subjects with a documented individual history of neck and/or upper extremity pain and/or functional/neurological deficit associated with the cervical level to be treated.
4. Subjects who are indicated for surgical treatment with the BEE® HA Cage with RESORBA® Synthetic Bone injectable bone substitute (RESORBA Medical GmbH).
5. Subjects who have completed at least 6 weeks of conservative non-operative treatment without obtaining adequate symptomatic relief.

Exclusion Criteria:

1. Subjects who have undergone previous spinal surgery either anterior or posterior.
2. Subjects with evidence of tumour and/or malignant disease with resultant life expectancy of less than two years.
3. Subjects with a known allergy to the material used in the instrumentation.
4. Subjects with evidence of an active infection and/or with any condition that would compromise their participation and follow-up in this clinical study.
5. Subjects who have known osteoporosis or severe osteopenia as determined by the Investigator.
6. Subjects who have any conditions outlined as contraindicated in the Instructions for Use.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospective study so patient population taken from those undergoing cervical spine fusion surgery.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) Questionnaire | 24 months
  Set of questions given to the subjects about experiencing pain during activities that are marked on a scale of 0-5 - whereby "0" is no pain and "5" is the worse pain. Maximum score for the questionnaire of "50" is possible.

CONTACTS AND LOCATIONS:
Locations (1):
- Bg Klinikum Bergmannstrost Halle, Halle, Germany

IPD SHARING:
Plan to Share IPD: No